CLINICAL TRIAL: NCT01267149
Title: Phase 4 Study - A Clinical Study Evaluaing the Efficacy, Safety, and Patient Satisfaction of Injectable Hylaronic Acid With 0.3% Lidocain Hydrochloride, Prevelle Silk, for Superficial, Vertical Perioral Lines and Superficial, Horizontal, Lateral Canthal Lines
Brief Title: A Clinical Study Evaluaing the Efficacy, Safety, and Patient Satisfaction of Injectable Hylaronic Acid With 0.3% Lidocain Hydrochloride, Prevelle Silk, for Superficial, Vertical Perioral Lines and Superficial, Horizontal, Lateral Canthal Lines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Mentor Worldwide, LLC (Industry)
Responsible Party: Mitchell Goldman MD, Goldman, Butterwick, Fitzpatrick and Groff
Other Study IDs: PRV-2010
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Wrinkles
Keywords: superficial vertical perioral lines; superficial horizontal and lateral canthal lines; correct moderate to severe facial wrinkles and folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Statistical Hypotheses The Null Hypothesis: There is no difference in the reduction of lines in the treated areas as compared to baseline.

Alternative Hypothesis: There is a difference in the reduction of lines in the treated areas as compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Females and males in good general health between 35 to 65 years of age.
* Must be willing to give and sign a HIPPA form, informed consent form and a photographic release form
* Patient is planning to undergo Prevelle Silk treatment
* A potential subject's must exhibit:

A. moderate to severe superficial, vertical perioral and horizontal canthus lines

* For FEMALE PATIENT OF CHILDBEARING POTENTIAL, must have had a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation) and is willing to use an acceptable form of birth control during the entire course of the study [i.e., acceptable methods of birth control are oral contraceptives, contraceptive patches/rings/implants Norplanit®, Depo-Provena®, double-barrier methods (e.g. condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the patient become sexually active]. All systemic birth control measures must be in consistent use at least 30 days prior to study participation
* Negative urine pregnancy test results at the time of study entry (if applicable)
* Must be willing to comply with study regimen and complete the entire course of the study.

Exclusion Criteria:

* A patient with any UNCONTROLLED systemic disease. A potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
* A patient with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* A patient with a known hypersensitivity to any of the components of the study medications
* A patient who is actively smoking or plans to smoke at any time of the duration of this study
* A patient with an active skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis, seborrheic dermatitis, herpes labialis)
* A patient planning any other cosmetic procedure to their facial area during the study period, other than the treatments that will be performed by the investigator
* A patient using any topical (prescription or over the counter) medicated creams, lotions, gels, balms, powders, etc. on the treatment areas during the study period
* A patient receiving any topical products containing alpha-hydroxy acids, salicylic acid, and vitamins C or D (includes derivatives thereof) on the perioral or lateral canthal areas within 7 days prior to or during the study period, other than the study products
* A patient receiving any investigational drug and/or has had a microdermabrasion (light or medium skin peel) treatment on their perioral or lateral canthal areas within 30 days prior to or during the study period
* A patient using any topical tretinoin product or derivative on their perioral or lateral canthal areas within 12 weeks prior to or during the study period
* A patient receiving a chemical peel, any systemic steroids, a non-ablative laser, light or radio frequency treatment and/or has had a Dermabrasion (deep skin peel) or ablative laser treatments on their perioral or lateral canthal areas must have discontinued the drug/treatment and/or had the procedure at least 6 months prior to entering the study
* A patient that has previously been treated with botulinum toxin in the perioral or lateral canthal areas within the past six months
* A patient that has previously been treated with dermal filler in the perioral or lateral canthal areas within the past year
* A patient that with a history of allergic reaction to a dermal filler or lidocaine
* A patient that with a history of a permanent filler to the perioral or lateral canthal areas
* A female patient who is pregnant, nursing an infant or planning a pregnancy during the study [throughout the course of the study, women of child-bearing potential must use reliable forms of contraception (i.e., oral contraceptive, intrauterine device, abstinence, or spermicides and condoms used in combination)]
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cosmetic Dermatology Practice Patients
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2010-08

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell P Goldman, MD, Principal Investigator — Dermatology and Cosmetic Laser Associated La Jolla
Locations (2):
- United States (2):
  - Goldman, Butterwick, Fitzpatrick and Groff, La Jolla, California
  - The Maas Clinic, San Francisco, California